CLINICAL TRIAL: NCT01743716
Title: Towards Identification of Genetic and Neural Predictors of Adolescent Depression
Brief Title: Genetic and Neural Predictors of Adolescent Depression
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Mclean Hospital (Other)
Collaborators: The Klingenstein Third Generation Foundation (Other); The Dana Foundation (Other)
Responsible Party: Principal Investigator, Randy P. Auerbach, Principal Investigator, Mclean Hospital
Other Study IDs: 2012P002351
Record Dates: First submitted 2012-12-04; First posted 2012-12-06 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; MDD; depression; adolescent
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Adolescent participants will provide a saliva sample for DNA analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- MDD Mothers: Adult women with a history of major depressive disorder (MDD) and a healthy adolescent daughter between the ages of 12-14
- Healthy Control Mothers: Adult women with no history of psychopathology and an adolescent daughter between the ages of 12-14
- High Risk Female Adolescents: Healthy female adolescents aged 12-14 with a mother in the MDD Mothers cohort
- Healthy Female Adolescents: Healthy female adolescents aged 12-14 with a mother in the Healthy Control Mothers cohort.

SUMMARY:
This study aims to examine the relationship between mood and brain activity in adolescent girls in order to better understand the genetic and neural predictors of adolescent depression. The participants in this study will be healthy female adolescents aged 12-14 and their mothers. They will participate for a total of six months. Adolescent participants will have three study sessions at McLean Hospital, and during two of them, their mothers will also have assessments. Adolescent assessments will include interviews, questionnaires, computer tasks, and collection of a saliva sample for genetic analyses. Their second study visit will include an fMRI scan. Parent assessments will include an interview, questionnaires, and a computer task.

ELIGIBILITY:
Adult Cohort

A. MDD Mothers Cohort Inclusion Criteria:

* Current or past Major Depressive Disorder
* English as first language or English fluency
* Biological daughter who meets inclusion/exclusion criteria for High Risk Female Adolescent

B. Healthy Control Mothers Cohort Inclusion Criteria:

* No history of psychopathology
* English as first language or English fluency
* Biological daughter who meets inclusion/exclusion criteria for Healthy Female Adolescent

Adolescent Cohort

General Inclusion Criteria for Adolescent Cohorts:

* Female
* Ages 12-14
* English as first language or English fluency
* Right handed

General Exclusion Criteria for Adolescent Cohorts:

* Past or present diagnosis of Major Depressive Disorder
* Past or present diagnosis of any anxiety disorder
* Past or present diagnosis of Bipolar Disorder
* Past or present diagnosis of ADHD
* Presence of medical or neurological illness (head injury, loss of consciousness greater than 5 minutes, seizure)
* Current use of psychotropic medication
* Presence of any contraindication for MRI:

  * Cardiac pacemakers
  * Metal clips on blood vessels (also called stents)
  * Artificial heart valve, artificial arms, hands, legs, etc.
  * Brain stimulator devices
  * Implanted drug pumps
  * Ear or eye implants
  * Known metal fragments in eyes
  * Exposure to metal filings or shrapnel (sheet metal workers, welders, and others)
  * Other metallic surgical hardware in vital area
  * Certain tattoos with metallic ink
  * Certain IUDs containing metal
  * Certain transdermal (skin) patches such as:
* NicoDerm (nicotine for tobacco dependence)
* Transderm Scop (scopolamine for motion sickness)
* Ortho Evra (birth control)

  * Positive urine pregnancy test

C. High Risk Female Adolescent Additional Inclusion Criterion:

• Biological daughter of participant in the MDD Mothers cohort

D. Healthy Female Adolescent Additional Inclusion Criterion:

• Biological daughter of participant in the Healthy Control Mothers cohort

Min Age: 12 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study will include two adult and two adolescent cohorts. The adult cohort includes two different groups of mothers: (a) MDD Mothers: Mothers with current or past major depressive disorder and (b) Healthy Control Mothers: Mothers with no history of psychopathology. The female adolescent cohorts are as follows: (c) High Risk Female Adolescents: Healthy female adolescents aged 12-14 with a mother reporting past or current MDD, (d) Healthy Female Adolescents: Healthy female adolescents aged 12-14 with a mother reporting no history of psychopathology.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-04 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Neurobiological Activity in Frontostriatal and Mesolimbic Regions | Baseline
Depressive Symptoms | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Randy P. Auerbach, PhD, Principal Investigator — Mclean Hospital; Diego A. Pizzagalli, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States